CLINICAL TRIAL: NCT04668625
Title: Risk of Infection of SARS-CoV-2 in a Massive Musical Show With Transmission Prevention Measures: Randomized Study
Brief Title: Risk of Infection of Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2), COVID-19, in a Massive Musical Show With Transmission Prevention Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Dr. Bonaventura Clotet Sala (Unknown); Dr. Josep Mª LLibre Codina (Unknown); Dr. Boris Revollo Barriga (Unknown); Dra. Lidia Ruiz Tabuenca (Unknown); Dr. Ignacio Blanco Guillermo (Unknown); Dra. Andrea Alemany Ortiz (Unknown); Dr. Roger Paredes Deiros (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRIMACOV
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: COVID-19 (SARS-CoV-2)
Keywords: SARS-CoV-2; COVID-19; Coronavirus; Superspreading event; Concert
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: All participants will be screened for a rapid Ag SARS-CoV-2 test detection. All negative subjects will be randomized to an experimental arm (participate in a massive musical event) or to a control arm (not participate in a massive musical event).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participate in a massive musical event
  Interventions: Behavioral: Participate in a massive musical event
- Control Group (No Intervention): Not participate in a massive musical event

INTERVENTIONS:
Behavioral: Participate in a massive musical event — Participate in a massive musical event
  Arms: Experimental group

SUMMARY:
The coronavirus disease 2019 (COVID-19) outbreak, caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), emerged in Wuhan in December 2019 and has spread globally, representing a serious threat to public health. While waiting for highly effective treatments or the development of an effective vaccine, it is necessary to reactivate key economic activities that are related to leisure and culture in an environment that is safest for the participants.

The use of a rapid screening test for SARS-CoV-2 viral antigens with high sensitivity could be a useful tool to detect asymptomatic SARS-CoV-2 infected people, and thus be able to carry out events related to leisure in a safe environment.

The aim of this study is to make a mass screening of asymptomatic infection of an (i) experimental group (public attending a massive mass musical show) and (ii) a control group (they will not enter the event) prior to entering to the event.

Randomization 1: 1 by random blocks of the participants with a negative antigen test in the experimental group (attending the event) and the control group (they will not enter the event).

Control with a new Polymerase Chain Reaction (PCR) test 8 days after the event (D8) in the participants of both randomized groups Control of the appearance of symptoms through a questionnaire 10 days after the event (D10), in the participants of both groups with a negative result on day 8.

Validation of a rapid antigen detection test by comparison with the PCR technique.

The indoor activity will include an array of measures designed to reducing the contagion risk, including: mandatory wearing a mask during the event, restricted outdoor areas of bar and smoking, enhanced ventilation of the whole indoor area, and avoiding queues.

All subjects will have downloaded an app in their smart phones to help contact and place tracing during the event, to trace potential transmissions. This app will remain active for 8 days, until the last virologic control.

The inclusion criteria will allow only subjects with an age <60 years, without comorbidities, and who do not live with old adults in their homes, to further reduce the risk of potential complications and transmission to at risk individuals.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) outbreak, caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), emerged in Wuhan in December 2019 and has spread globally, representing a serious threat to public health. While 80% of patients are asymptomatic or have a mild illness, 20% develop a severe illness. The predominant symptoms include fever, cough, and myalgia. Mild disease can resolve without medical attention or it can progress to pneumonia and respiratory failure requiring hospitalization. Patients can rapidly progress to acute respiratory distress syndrome (ARDS) with multiple organ dysfunction and death.

The degree to which the virus is infectious during the incubation period is uncertain, but it has been shown that the pharynx reaches peak viral load before day 5, and this peak viral load is 1,000 times higher than in severe acute respiratory syndrome coronavirus (SARS-CoV). This active and high viral clearance from the pharynx at a time when symptoms are still mild makes the transmission of SARS-CoV-2 more efficient than that of SARS-CoV. Later in the disease, COVID-19 resembles SARS in terms of replication in the lower respiratory tract. The decrease in viral load appears to be slow, and there is no sudden shedding of the virus at the time of seroconversion. Seroconversion, at the beginning of week 2, has been observed to coincide with a slow but steady decrease in sputum viral load. Prolonged viral shedding in sputum is relevant not only for infection control in hospitals and discharge management, but also for asymptomatic people who can transmit the virus for longer periods after infection.

Although it is true that the majority of people infected by SARS-CoV-2 will have a benign course with few symptoms, approximately 20% will require hospitalization and 5% will present serious complications and admission to an intensive care unit, this is it translates into a saturation and collapse of health systems, with a high percentage of mortality in relation to it. Unprecedented confinement measures have been implemented that have been effective in containing the progression of the number of infections, but these have had a great social and economic impact, among others with a paralysis of most of the activities related to leisure (concerts , music festivals, theaters, etc.) that are an important component in the economy of most of the countries of the European community. While waiting for highly effective treatments or the development of an effective vaccine, it is necessary to reactivate key economic activities that are related to leisure and culture in an environment that is safest for the participants.

The use of a rapid screening test for SARS-CoV-2 viral antigens with high sensitivity could be a useful tool to detect asymptomatic SARS-CoV-2 infected people, and thus be able to carry out events related to leisure in a safe environment.

It is necessary to implement versatile circuits in which diagnoses with rapid tests can be carried out in the same place of the events in a massive way and to be able to communicate the results of the tests to the assistants at the same time, in order to do this screening of people that they give negative and carry out activities with them in a safe environment for all participants.

The aim of this study is to make a mass screening of asymptomatic infection of an (i) experimental group (public attending a massive mass musical show) and (ii) a control group (they will not enter the event) prior to entering to the event.

Randomization 1: 1 by random blocks of the participants with a negative antigen test in the experimental group (attending the event) and the control group (they will not enter the event).

Control with a new PCR test 8 days after the event (D8) in the participants of both randomized groups Control of the appearance of symptoms through a questionnaire 10 days after the event (D10), in the participants of both groups with a negative result on day 8.

Validation of a rapid antigen detection test by comparison with the PCR technique.

The indoor activity will include an array of measures designed to reducing the contagion risk, including: mandatory wearing a mask during the event, restricted outdoor areas of bar and smoking, enhanced ventilation of the whole indoor area, and avoiding queues.

All subjects will have downloaded an app in their smart phones to help contact and place tracing during the event, to trace potential transmissions. This app will remain active for 8 days, until the last virologic control.

The inclusion criteria will allow only subjects with an age <60 years, without comorbidities, and who do not live with old adults in their homes, to further reduce the risk of potential complications and transmission to at risk individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18-59 years) with interest to attend the scheduled musical event who agree to participate in the study after signing the informed consent, including explicit acceptance of the measures implemented to reduce the risk of transmission of SARS-CoV-2.
* Negative antigen test performed up to 24 h before the event, in nasopharyngeal swab.

Exclusion Criteria:

* Hypertension
* Diabetes Mellitus.
* Ischemic heart disease.
* Any type of Cancer in active treatment.
* Chronic lung diseases such as chronic obstructive pulmonary disease (COPD) and asthma.
* Have a positive test for detection of SARS-CoV-2 by the rapid antigen test
* Who have a body temperature higher than 37.0º on the same day of the event
* Who have a confirmed diagnosis for SARS-CoV-2 in the two weeks prior to the event
* Report any symptoms suggestive of a SARS-CoV-2 infection in the 10 days prior to the study
* Who have been in contact with a person with a confirmed diagnosis of SARS-CoV-2 infection within two weeks prior to the event.
* Living with a person over 70 years of age (inclusive).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Incidence rate of people infected with SARS-CoV-2 8 days after randomization | At 8 days
  Incidence rate of people infected with SARS-CoV-2 8 days after randomization, detected by PCR in nasopharyngeal aspirate, on the experimental and the control group.

SECONDARY OUTCOMES:
SARS-CoV-2 genome sequence | At 8 days
  Nasopharyngeal swab samples will be stored in case SARS-CoV-2 infections are documented for sequencing purposes to assess the possibility of spreading clusters during the event. Data will be matched with a Global Positioning System (GPS) smart phone tracking localization during the concert.
Incidence rate of appearance of symptoms compatible with COVID 19 | At 10 days
  Incidence rate of appearance of symptoms compatible with COVID 19 in those attending the event after 10 days (D10).
Time spent in testing the total number of participants in the study. | At day 0
  Time spent in testing the total number of participants in the study.
Comparison of the diagnostic sensitivity of rapid antigen tests for SARS-CoV-2 compared to PCR in asymptomatic subjects. | At day 0
  We will compare the diagnostic sensitivity of rapid antigen tests for SARS-CoV-2 compared to PCR in asymptomatic subjects.
Comparison of the diagnostic sensitivity of rapid antigen tests for SARS-CoV-2 using a nasopharyngeal swab sample compared to sample obtained trough saliva | At day 0
  We will compare the diagnostic sensitivity of rapid antigen tests for SARS-CoV-2 using a nasopharyngeal swab sample compared to sample obtained trough saliva, in positive cases by this technique.
Presence of viable SARS-CoV-2 from cell culture | At day 0
  Presence of viable SARS-CoV-2 from cell culture in all cases with negative Ag and positive PCR.
Satisfaction in relation to the test procedure | At 10 days
  Assessment of the results obtained on satisfaction in relation to the test procedure of those attending the event through a questionnaire.
  Questions:
  1. I have had all the necessary prior information to participate in this study
  2. I have felt properly cared for by the health personnel
  3. I have felt properly cared for by the room staff
  4. I have behaved naturally without feeling conditioned by the measures of the protocol during the event
  5. I have been able to enjoy the performance in a satisfactory way
  6. I will attend other leisure events in closed spaces following this same protocol
  It can be answered with a scale from 0 to 10 (0 not satisfied at all, 10 extremely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet Sala, PhD, MD, Principal Investigator — Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia; Boris Revollo Barriga, PhD, MD, Principal Investigator — Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia; Josep Mª LLIBRRE CODINA, PhD, MD, Principal Investigator — Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Revollo B, Blanco I, Soler P, Toro J, Izquierdo-Useros N, Puig J, Puig X, Navarro-Perez V, Casan C, Ruiz L, Perez-Zsolt D, Videla S, Clotet B, Llibre JM. Same-day SARS-CoV-2 antigen test screening in an indoor mass-gathering live music event: a randomised controlled trial. Lancet Infect Dis. 2021 Oct;21(10):1365-1372. doi: 10.1016/S1473-3099(21)00268-1. Epub 2021 May 27. PMID 34051886